CLINICAL TRIAL: NCT03013764
Title: Interaction Between Diet Composition and Physical Inactivity on Insulin Sensitivity and β-cell Function
Brief Title: Diet Composition and Physical Inactivity on Insulin Sensitivity and β-cell Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: American Egg Board - 00050021
Record Dates: First submitted 2016-12-20; First posted 2017-01-06 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Physical Inactivity; Dietary Protein
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal protein intake (Placebo Comparator): subjects will undergo 10 days of low physical activity while consuming a normal protein diet
  Interventions: Behavioral: normal protein diet
- high protein intake (Experimental): subjects will undergo 10 days of low physical activity while consuming a high protein diet
  Interventions: Behavioral: high protein intake

INTERVENTIONS:
Behavioral: normal protein diet — subjects will undergo 10 days of low physical activity while consuming a normal protein diet
  Arms: normal protein intake
Behavioral: high protein intake — subjects will undergo 10 days of low physical activity while consuming a high protein diet
  Arms: high protein intake

SUMMARY:
Physical inactivity results in reductions in glucose tolerance and less sensitivity to insulin. If this inactivity lasts long enough it can result in insulin resistance and type 2 diabetes. A high protein diet can reduce elevated glucose levels in individuals with type 2 diabetes. Thus the investigators are interested in establishing if during a period of inactivity if a diet modification can minimize the glucose changes normally observed with inactivity. The objective of this project is to determine if short-term high protein (HP) feeding protects against the changes in glucose levels normally observed with physical inactivity. The investigators will also examine measures of blood vessel function, blood lipid and blood pressure.

Twelve subjects will complete two 10 day study periods of reduced physical activity and will be studied before and after each of these study periods. For their testing subjects will have the following measurements: postprandial glucose responses to a mixed meal, 24 h free living blood pressure control during acute physical inactivity, blood lipids, changes in body composition, changes in circadian rhythm using skin temperature (ibutton), measurement of aerobic capacity (VO2 max), blood vessel responsiveness (flow mediated dilation -FMD) and changes in free living glucose levels (continuous glucose monitoring system (CGMS). Subjects will complete two conditions (high protein -HP vs normal protein - NP diets) in a randomized cross-over design. In the inactive phase subjects will reduce there steps to <5,000 steps/d while consuming either a HP or NP diet. Completion of the study will take 8-10 weeks.

DETAILED DESCRIPTION:
It is well known that insulin resistance increases the risk of cardiovascular disease and type 2 diabetes, which substantially impact mortality and morbidity and presents a significant economic burden. Energy restriction with or without exercise has been demonstrated to attenuate/reverse the development of insulin resistance and reduce the risk of cardiovascular disease and type 2 diabetes. Indeed, accumulating evidence suggests that diets high in protein may possess additional protection against the development of insulin resistance during energy restriction. Layman et al. found that a high protein diet (HP) (PRO 125 g/d) compared with an isocaloric high carbohydrate diet (HCHO) (PRO 68 g/d) resulted in greater reductions in fasting glucose and 2 h postprandial insulin levels during 16 weeks of energy restriction in overweight women. Similarly, a hypocaloric high protein diet (PRO 45% vs 20%; 21 d diet treatment) increased glucose oxidation and improved insulin sensitivity compared to an isocaloric high carbohydrate diet during a euglycemic hyperinsulinemic clamp procedure. In addition, markers of inflammation, β-cell function, and postprandial glucose and insulin levels were improved in addition to increased resting energy expenditure after 6 months of hypocaloric HP compared with HCHO diet in premenopausal women independent of weight loss. The increase in REE and improvement in adipose tissue function may be a potential mechanism by which HP diet improves β-cell function since NEFAs are lower, which may reduce lipotoxicity on the pancreas.

It is evident that physical inactivity (highlighted from bed rest studies) impairs glucose tolerance, insulin sensitivity, vascular function, and muscle protein synthesis in both healthy and obese individuals. This model of inactivity, however, is extreme and does not recapitulate the physical inactivity paradigm seen in the natural human environment. Consequently, a less extreme reduction in daily physical activity (>10,000 steps/d to ~1,500 steps/d) results in significant reductions in insulin sensitivity, glucose tolerance, and insulin-stimulated muscle Akt phosphorylation, suggesting that the impairments in insulin sensitivity and glucose tolerance precede changes in body composition. A reduction in ambulatory activity is a highly valid and translatable model to study the role of inactivity on the development of metabolic disease, as most individuals go through periods of inactivity, and it has been shown that a reduction in daily steps decreases insulin sensitivity and increases visceral adiposity. To date, no study has tested the effects of diet composition on the perturbations of physical inactivity. It is important to know if increasing protein intake mitigates the negative perturbations of reduced ambulatory activity.

Thus, the overall objective of this project is to determine the extent to which short-term high protein (HP) feeding may protect against the metabolic perturbations of physical inactivity (i.e. PPG, hyperinsulinemia, and insulin sensitivity). The investigators will also examine measures of vascular function and free living blood pressure in addition to lipemic responses (i.e. FFAs, triglycerides, cholesterol, and lipoproteins) to determine if HP diet impacts vascular function and lipemic responses during short term physical inactivity.

Trial Objectives and Purpose

The specific aims of this project include the following:

Specific Aim 1: To determine if HP diet during a period of low physical activity will lower the insulin response to a meal, and help to maintain insulin sensitivity and β-cell function during a laboratory based mixed meal test (MMT) with stable isotope tracers.

Specific Aim 2: To determine if a HP diet during a period of low physical activity will maintain glycemic control measured by continuous glucose monitoring (CGM) in healthy, recreationally active, young individuals.

ELIGIBILITY:
Inclusion Criteria:

1. BMI <28 kg/m2
2. No known cardiovascular, kidney, or liver disease.
3. No history of surgery for weight loss and weight stable for prior 3 months (weight change < 3 kg).
4. Physically active individual (90 minutes of primarily whole body aerobic physical activity <3 days per week and taking greater than 10,000 steps per day)
5. Between 18-45 yr of age.
6. Participants who consume on average less than 18% of total calories as protein

Exclusion Criteria:

1. History of alcohol use (< 20 g/day for males and > 10 g/day for females)
2. Smoker.
3. BMI < 28 kg/m2
4. Kidney or liver disease.
5. Physically inactive (completing < 75 min of whole body aerobic activity <3 times per week or obtaining <10,000 steps/day)
6. Pregnant or lactating
7. <18 or >45 yr of age
8. High protein consumers (>20% of total daily calories as protein)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
glucose excursions | change in from baseline

SECONDARY OUTCOMES:
insulin sensitivity | change in from baseline
blood lipids | change in from baseline
insulin, FFA and other hormones (e.g. glucagon, adropin, etc) | change in from baseline
endothelial function | change in from baseline
beta cell function | change in from baseline

CONTACTS AND LOCATIONS:
Overall Officials: jill kanaley, Phd, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winn NC, Pettit-Mee R, Walsh LK, Restaino RM, Ready ST, Padilla J, Kanaley JA. Metabolic Implications of Diet and Energy Intake during Physical Inactivity. Med Sci Sports Exerc. 2019 May;51(5):995-1005. doi: 10.1249/MSS.0000000000001892. PMID 30694977